CLINICAL TRIAL: NCT04094415
Title: SURE ITALY: A Multi-centre, Prospective, Non-interventional Study Investigating the Effectiveness of Once-weekly Subcutaneous Semaglutide in a Real World Adult Population With Type 2 Diabetes
Brief Title: A Research Study Looking at How Semaglutide Works in People With Type 2 Diabetes in Italy, as Part of Local Clinical Practice
Acronym: SURE ITALY
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-4549; U1111-1233-2023 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semaglutide: Participants will receive semaglutide at the treating physician's discretion as part of the usual clinical practice. The prescription and use of semaglutide is completely independent of this study. Total study duration for the individual patient will be approximately 30 weeks.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Patients will be treated with commercially available semaglutide in a prefilled pen injector (FlexTouch® variant) according to routine local clinical practice at the discretion of the treating physician. Other anti-hyperglycaemic treatments will be prescribed at the physician's discretion.The decision to initiate treatment with semaglutide is at the treating physician's discretion, and clearly separated from the decision to include the patient in the study.

SUMMARY:
The purpose of the study is to collect information on how semaglutide works in real world patients. Participants will get semaglutide prescribed to them by their doctor. The study will last for about 6 to 8 months. Participants will be asked to complete some questionnaires about their health and your diabetes treatment. Participants will complete these during their normally scheduled visits with their doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* The decision to initiate treatment with commercially available semaglutide has been made by the patient/Legally Acceptable Representative and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age 18 years or older at the time of signing informed consent
* Diagnosed with type 2 diabetes at least 12 weeks prior to inclusion
* Available and documented haemoglobin A1c (HbA1c) value equal to or less than 12 weeks prior to initiation of semaglutide treatment

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Treatment with any investigational drug within 90 days prior to enrolment into the study
* Hypersensitivity to semaglutide or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin A1c (HbA1c) (measured in percent) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Measured in % points
Change in HbA1c (measured in mmol/mol) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Measured in mmol/mol

SECONDARY OUTCOMES:
Change in body weight (measured in kg) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Measured in kg
Change in body weight (measured in percent) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Measured in %
Change in waist circumference | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Measured in cm
HbA1c level at end of study: below 8.0% (64 mmol/mol) (yes/no) | At end of study (week 28 to 38)
  Number of participants who achieved/not achieved HbA1c level at end of study: below 8.0%
HbA1c level at end of study: below 7.5% (59 mmol/mol) (yes/no) | At end of study (week 28 to 38)
  Number of participants who achieved/not achieved HbA1c level at end of study: below 7.5%
HbA1c level at end of study: below 7.0% (53 mmol/mol) (yes/no) | At end of study (week 28 to 38)
  Number of participants who achieved/not achieved HbA1c level at end of study: below 7.0%
Reduction in HbA1c from baseline to end of study of 1.0% point or more (Y/N) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Number of participants who achieved/not achieved reduction in HbA1c of 1.0% point or more
Weight reduction of 3.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Number of participants who achieved/not achieved weight reduction of 3.0% or more
Weight reduction of 5.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Number of participants who achieved/not achieved weight reduction of 5.0% or more
HbA1c reduction of 1.0% point or more and weight reduction of 3.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28 to 38)
  Number of participants who achieved/not achieved HbA1c reduction of 1.0% point or more and weight reduction of 3.0% or more
Patient reported severe or documented hypoglycaemia (yes/no) | Between baseline (week 0) and end of study (week 28-38)
  Number of patients who reported/not reported severe or documented hypoglycaemia
Change in score for Diabetes Treatment Satisfaction Questionnaire - Status (DTSQs) (absolute treatment satisfaction): Total treatment satisfaction | Baseline (week 0), end of study (week 28 to 38)
  The status version (DTSQs) provides a measure of how satisfied patients are with their current diabetes treatment. It consists of 8 questions, which are to be answered on a Likert scale from 0 to 6 (0 = very dissatisfied to 6 = very satisfied). Six questions are summed to produce a total Treatment Satisfaction score. The remaining two questions are concerning perceived frequency of hyperglycaemia and perceived frequency of hypoglycaemia, respectively.
Change in score for Diabetes Treatment Satisfaction Questionnaire - Change (DTSQc) (relative treatment satisfaction): Total treatment satisfaction ) | Baseline (week 0), end of study (week 28 to 38
  The change version (DTSQc) has the same 8 items as the status version, but is reworded to direct the patients to compare the experience of the current treatment with the experience of previous treatment. Each question is scored on a scale of -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change.
Change in score for Short Form (SF)-36 v2: Physical summary component | Baseline (week 0), end of study (week 28 to 38)
  The SF-36®v2 questionnaire has 36 questions grouped into eight domains termed: physical functioning, bodily pain, role-physical, general health, vitality, social functioning, role-emotional and mental health, which again can be combined to give two summary component scores (overall mental- and physical health).
Change in score for SF-36 v2: Mental summary component | Baseline (week 0), end of study (week 28 to 38)
  The SF-36®v2 questionnaire has 36 questions grouped into eight domains termed: physical functioning, bodily pain, role-physical, general health, vitality, social functioning, role-emotional and mental health, which again can be combined to give two summary component scores (overall mental- and physical health).
Patient completed the study under treatment with semaglutide (yes/no) | At end of study (week 28 to 38)
  Number of patients who completed/not completed the study under treatment with semaglutide

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (31):
- Italy (31):
  - Novo Nordisk Investigational Site, Bagno a Ripoli
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Brindisi
  - Novo Nordisk Investigational Site, Casarano (Lecce)
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieri Torino
  - Novo Nordisk Investigational Site, Cipolleto Perugia
  - Novo Nordisk Investigational Site, Foggia
  - Novo Nordisk Investigational Site, Gaeta
  - Novo Nordisk Investigational Site, Genova
  - Novo Nordisk Investigational Site, Livorno
  - Novo Nordisk Investigational Site, L’Aquila
  - Novo Nordisk Investigational Site, Macerata
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Negrar (VR)
  - Novo Nordisk Investigational Site, Orbassano
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Prato
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Rome
  - Novo Nordisk Investigational Site, Rozzano (MI)
  - Novo Nordisk Investigational Site, Sesto San Giovanni (MI)
  - Novo Nordisk Investigational Site, Treviglio (Bergamo)
  - Novo Nordisk Investigational Site, Treviso
  - Novo Nordisk Investigational Site, Udine
  - Novo Nordisk Investigational Site, Vicenza
  - Novo Nordisk Investigational Site, Vigevano

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Background] Napoli R, Berra C, Catarig AM, Di Loreto C, Donatiello E, Berentzen TL, Pitocco D, Giorgino F. Once-weekly semaglutide use in patients with type 2 diabetes: Real-world data from the SURE Italy observational study. Diabetes Obes Metab. 2023 Jun;25(6):1658-1667. doi: 10.1111/dom.15020. Epub 2023 Mar 12. PMID 36789682